CLINICAL TRIAL: NCT00440999
Title: A Phase III Comparative (Double-blind, Double-dummy) Randomised Multicentre Study to Assess the Safety & Efficacy of Oral Pyronaridine Artesunate (180:60 mg) Versus Chloroquine (155 mg) in Children & Adult Patients With Acute Vivax Malaria
Brief Title: Pyronaridine Artesunate (3:1) in Children and Adults With Acute Plasmodium Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-C-006-06
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: P vivax; malaria; artemisinin based combination therapy (ACT); antimalarial; pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Chloroquine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pyronaridine artesunate (Experimental): The tablet strength is 180:60 mg oral PA plus chloroquine-placebo. Depending on their body weight, patients receive 1 to 4 tablets once a day, for 3 days. The actual dose-level range covered by this regimen is 7.2: 2.4 mg/kg to 13.8:4.6 mg/kg pyronaridine artesunate.
  Interventions: Drug: Pyronaridine artesunate
- chloroquine (Active Comparator): The tablet strength is 155 mg oral chloroquine plus PA-placebo.
  Patients receive:
  For adults: 620 mg (i.e. 4 tablets) on Days 0 and 1 and 310 mg (i.e. 2 tablets) on Day 2. For children: 10 mg/kg on Days 0 and 1 and 5 mg/kg on Day 2.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Pyronaridine artesunate
  Other Names: Pyramax
  Arms: pyronaridine artesunate
Drug: Chloroquine
  Arms: chloroquine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the fixed combination of pyronaridine artesunate (Pyramax®, PA) (180:60 mg) with that of standard chloroquine therapy in children and adults with acute, uncomplicated Plasmodium vivax malaria.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, double-blind, double-dummy, parallel-group, non-inferiority study comparing the efficacy and safety of the fixed combination of pyronaridine/artesunate (ie, PP/AS [PA]) (180:60 mg) with that of standard chloroquine therapy in children and adults with acute uncomplicated P. vivax malaria. The study population will include 456 patients, comprising male and female children (≥20 kg body weight) and adults recruited from study sites in South East Asia and India.

Patients will be randomised in a 1:1 ratio to receive either oral PA (180:60 mg tablets) plus chloroquine-placebo or oral chloroquine (155 mg tablets).plus PA-placebo, once a day for 3 consecutive days (Days 0, 1, and 2). For PA, posology was based on body weight ranges with subjects receiving 1 to 4 tablets depending on their body weight. The dose range covered by this regimen is 7.2:2.4 mg/kg to 13.8:4.6 mg/kg, which has been shown to be effective and safe in Phase I and II studies. The chloroquine daily dose is 10 mg/kg on Days 0 and 1 and 5 mg/kg on Day 2 for children, and 620 mg on Days 0 and 1 and 310 mg on Day 2 for adults.

Patients will be confined to the study facility for ≥4 days (Days 0,1,2 & 3) and ideally remain near the study site for ≥7 days, or once fever and parasite clearance has been confirmed for ≥24 hours - whichever occurs later.

The primary efficacy end point for the study is the crude cure rate on Day 14, which is defined as the absence of P. vivax parasitaemia on Day 14. Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

For patients who complete the study up to Day 28 and who have normal glucose-6-phosphate dehydrogenase (G-6-PD) activity, a 14-day course of primaquine (15 mg/day for adults and 0.3 mg/kg/day for children) will be administered starting on Day 28 to complete their radical cure. Subjects who are deficient in G-6-PD and who completed the study up to Day 28 will be treated per country policy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 3 and 60 years, inclusive.
2. Body weight between 20 kg and 90 kg with no clinical evidence of severe malnutrition.
3. Presence of acute uncomplicated P. vivax mono-infection confirmed by:

   * Fever, as defined by axillary/tympanic temperature ≥37.5°C or oral/rectal temperature ≥38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   * Positive microscopy of P. vivax with parasite density ≥250/ mcL of blood (including at least 50% of asexual parasites).
4. Written informed consent, in accordance with local practice, provided by patient and/or parent/guardian/spouse. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations.
5. Ability to swallow oral medication.
6. Ability and willingness to participate based on information given to patient or parent or guardian and access to health facility.

Exclusion Criteria:

1. Presence of a mixed Plasmodium infection.
2. Presence of other clinical condition requiring hospitalization.
3. Presence of significant anaemia, as defined by Hb <8 g/dL.
4. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTc interval ≥450 msec), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including recent head trauma).
5. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine, chloroquine or artesunate or other artemisinins.
6. Known history of hypersensitivity, allergic or adverse reactions to chloroquine, primaquine and related agents.
7. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab).
8. Known seropositive HIV antibody.
9. Have received any antimalarial treatment in the preceding 2 weeks, as determined by history and, whenever feasible, by screening test.
10. Have received antibacterial with known antimalarial activity in the preceding 2 weeks.
11. Have received any investigational drug within the past 4 weeks.
12. Liver function tests (AST/ALT levels) >2.5 times the upper limit of normal range.
13. Known significant renal impairment as indicated by serum creatinine levels of >1.4 mg/dL.
14. Female patients of child-bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures to not become pregnant during the study period.
15. Previous participation in the present clinical trial with PA.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 456 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Borghini Fuhrer, PhD, Study Director — Medicines for Malaria Venture
Locations (5):
- Pailin Referral Hospital, Pailin, Pailin, Cambodia
- Wentlock District Hospital, Mangalore, India
- RSUD TC Hillers, Maumere, Nusa Tenggara Timur, Indonesia
- Thailand (2):
  - MaeLamad District Hospital, Mae Ramat, Changwat Tak
  - MaeSod General Hospital, Mae Sot, Changwat Tak

REFERENCES:
- [Result] Poravuth Y, Socheat D, Rueangweerayut R, Uthaisin C, Pyae Phyo A, Valecha N, Rao BH, Tjitra E, Purnama A, Borghini-Fuhrer I, Duparc S, Shin CS, Fleckenstein L. Pyronaridine-artesunate versus chloroquine in patients with acute Plasmodium vivax malaria: a randomized, double-blind, non-inferiority trial. PLoS One. 2011 Jan 18;6(1):e14501. doi: 10.1371/journal.pone.0014501. PMID 21267072
- [Derived] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102

RESULTS

PARTICIPANT FLOW:
Groups:
- Pyronaridine - Artesunate: Subjects receive oral active-pyronaridine artesunate (tablet 180:60 mg) + chloroquine-placebo, once a day for 3 consecutive days (D0, 1, and 2).
  Posology was based on body weight ranges with subjects receiving 1 to 4 tablets depending on their body weight. The actual dose range covered by this regimen was 7.2:2.4 mg/kg to 13.8:4.6 mg/kg.
- Chloroquine: Subjects receive oral active-chloroquine (tablet 155 mg) + pyronaridine artesunate - placebo, once per day for 3 consecutive days (D0, 1, and 2).
  The daily dose is 10 mg/kg on Days 0 and 1, and 5 mg/kg on Day 2 for children, and 620 mg on Days 0 and 1, and 310 mg on Day 2 for adults.
Period: Overall Study
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Started | 228 | 228
Completed | 193 | 187
Not Completed | 35 | 41
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 6 | 7
Not completed — Lost to Follow-up | 19 | 12
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Subjets missed the visit | 1 | 0
Not completed — Mixed infection at entry | 1 | 0
Not completed — P. falciparum malaria | 5 | 14
Not completed — Subj left hosp without inform staff | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population, defined as all randomized subjects who received any amount of study medication. Males/Females between ages of 3 and 60 years, with body weight ≥ 20 kg.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyronaridine - Artesunate | Chloroquine | Total
Number analyzed (Participants) | 228 | 228 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects total and per country/site
  years
    Total | 27.0 (11.7) | 26.4 (10.93) | 26.7 (11.04)
    Cambodia: number analyzed (Participants) | 77 | 77 | 154
    Cambodia | 21.0 (8.93) | 23.0 (9.92) | 22.0 (9.46)
    India: number analyzed (Participants) | 39 | 41 | 80
    India | 31.5 (12.20) | 27.9 (11.99) | 29.7 (12.15)
    Indonesia/Maumere: number analyzed (Participants) | 13 | 11 | 24
    Indonesia/Maumere | 26.7 (10.59) | 18.6 (9.07) | 23.0 (10.54)
    Thailand/Mae Sot: number analyzed (Participants) | 49 | 50 | 99
    Thailand/Mae Sot | 29.6 (11.15) | 29.6 (9.80) | 29.6 (10.44)
    Thailand/Mae Ramat: number analyzed (Participants) | 50 | 49 | 99
    Thailand/Mae Ramat | 30.5 (9.93) | 29.0 (11.04) | 29.7 (10.47)
Age, Customized [Count of Participants; unit: Participants]
  ≤12 years | 14 | 13 | 27
  >12 years | 214 | 215 | 429
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects total and per country/site
  Participants
    Total: Female | 56 | 64 | 120
    Total: Male | 172 | 164 | 336
    Cambodia: number analyzed (Participants) | 77 | 77 | 154
    Cambodia: Female | 25 | 27 | 52
    Cambodia: Male | 52 | 50 | 102
    India: number analyzed (Participants) | 39 | 41 | 80
    India: Female | 5 | 7 | 12
    India: Male | 34 | 34 | 68
    Indonesia/Maumere: number analyzed (Participants) | 13 | 11 | 24
    Indonesia/Maumere: Female | 6 | 3 | 9
    Indonesia/Maumere: Male | 7 | 8 | 15
    Thailand/Mae Sot: number analyzed (Participants) | 49 | 50 | 99
    Thailand/Mae Sot: Female | 11 | 11 | 22
    Thailand/Mae Sot: Male | 38 | 39 | 77
    Thailand/Mae Ramat: number analyzed (Participants) | 50 | 49 | 99
    Thailand/Mae Ramat: Female | 9 | 16 | 25
    Thailand/Mae Ramat: Male | 41 | 33 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 228 | 228 | 456
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Cambodia | 77 | 77 | 154
  Thailand | 99 | 99 | 198
  India | 39 | 41 | 80
  Indonesia | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Crude Cure Rate on Day 14
Description: Cure rate on Day 14 is defined as the absence of P. vivax parasitaemia on Day 14 irrespective of temperature (axillary, oral, tympanic, rectal) without previously meeting any of the criteria of treatment failure throughout the follow-up period.
Time Frame: Day 14
Population: Efficacy evaluable population: completed a full course of study medication, did not miss a dose, did not use a concomitant medication that may have interfered with the treatment outcome up to D14, did not have a concomitant disease which may have interfered with the classification of the treatment outcome, did not have major protocol deviations.
Measure: Count of Participants; unit: Participants
Groups:
- Pyronaridine Artesunate: Subjects receive oral active-pyronaridine artesunate (tablet 180:60 mg) + chloroquine-placebo, once a day for 3 consecutive days (Day 0, 1, and 2).
  Posology was based on body weight ranges with subjects receiving 1 to 4 tablets depending on their body weight. The actual dose range covered by this regimen was 7.2:2.4 mg/kg to 13.8:4.6 mg/kg.
- Chloroquine: Subjects receive oral active-chloroquine (tablet 155 mg) + pyronaridine artesunate - placebo, once per day for 3 consecutive days (Day 0, 1, and 2).
  The daily dose is 10 mg/kg on Days 0 and 1, and 5 mg/kg on Day 2 for children, and 620 mg on Days 0 and 1, and 310 mg on Day 2 for adults.
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 218 | 209
Participants
  Total cured | 217 | 209
  Cambodia: number analyzed (Participants) | 75 | 73
  Cambodia | 75 | 73
  India: number analyzed (Participants) | 33 | 33
  India | 33 | 33
  Indonesia/Maumere: number analyzed (Participants) | 11 | 10
  Indonesia/Maumere | 11 | 10
  Thailand/Mae Sot: number analyzed (Participants) | 49 | 46
  Thailand/Mae Sot | 49 | 46
  Thailand/Mae Ramat: number analyzed (Participants) | 50 | 47
  Thailand/Mae Ramat | 50 | 47
  baseline P. vivax = 250-5,000/uL: number analyzed (Participants) | 70 | 80
  baseline P. vivax = 250-5,000/uL | 69 | 80
  baseline P. vivax = >5,000/uL-10,000/uL: number analyzed (Participants) | 58 | 59
  baseline P. vivax = >5,000/uL-10,000/uL | 58 | 59
  baseline P. vivax = >10,000/uL: number analyzed (Participants) | 89 | 70
  baseline P. vivax = >10,000/uL | 89 | 70
  age ≤ 12 years: number analyzed (Participants) | 13 | 11
  age ≤ 12 years | 13 | 11
  age ≥ 12 years: number analyzed (Participants) | 205 | 198
  age ≥ 12 years | 204 | 198
  Gender - Male: number analyzed (Participants) | 164 | 148
  Gender - Male | 164 | 148
  Gender - Female: number analyzed (Participants) | 54 | 61
  Gender - Female | 53 | 61
  Previous P. vivax episode in the past = no: number analyzed (Participants) | 107 | 93
  Previous P. vivax episode in the past = no | 107 | 93
  Previous P. vivax episode in the past = yes: number analyzed (Participants) | 111 | 116
  Previous P. vivax episode in the past = yes | 110 | 116
Statistical Analysis 1: Comparison: Pyronaridine Artesunate vs Chloroquine; Null hypothesis: The cure rate on Day 14 for the PA group is inferior to the cure rate on Day 14 for the chloroquine group by more than 10%. Was tested against the alternative: Alternative hypothesis: The cure rate on Day 14 for the PA group was not inferior to the cure rate on Day 14 for the chloroquine group by more than 10%; Test type: Non-Inferiority — The primary efficacy analysis tested the non-inferiority of the PA group compared to the comparator group with regard to the crude cure rate on Day 14 using the 2-sided 95% confidence interval (CI) (Newcombe-Wilson score method without continuity correction) and a 10% non-inferiority margin. Non-inferiority was claimed if the lower limit of the 2-sided 95% CI for the difference in cure rates on Day 14 was >10%; Difference in cure rate = -0.5, 95% CI 2-sided [-2.6 to 1.4] — Conclusion: non-inferiority between PA & chloroquine

2. Secondary Outcome: Crude Cure Rate on Days 21 and 28.
Description: Cure on Day 21 and 28 is defined as the absence of P. vivax parasitaemia on Day 21 and 28 irrespective of temperature (axillary, oral, tympanic, rectal) without previously meeting any of the criteria of treatment failure throughout the follow-up period.
Time Frame: Day 21 and 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of cured subjects
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 218 | 209
percentage of cured subjects
  Cure rate (%) at Day 21: number analyzed (Participants) | 214 | 202
  Cure rate (%) at Day 21 | 99.5 [97.4 to 100.0] | 99.5 [97.3 to 100.0]
  Cure rate (%) at Day 28: number analyzed (Participants) | 208 | 196
  Cure rate (%) at Day 28 | 97.1 [93.8 to 98.9] | 98.0 [94.9 to 99.4]

3. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time is defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance is defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart.
Time Frame: Days 0 to 42
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 218 | 209
hours | 23.1 [16.3 to 23.5] | 32.0 [31.7 to 32.0]

4. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time is defined as the time from first dosing to the first normal reading of temperature (<37.5°C for axillary/tympanic or <38°C for oral/rectal) for 2 consecutive normal temperature readings taken between 7 and 25 hours apart.
Time Frame: Days 0 to 42
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 168 | 154
hours | 15.8 [15.5 to 16.0] | 23.8 [16.0 to 24.0]

5. Secondary Outcome: Percentage of Subjects With Parasite Clearance on Days 1, 2, and 3
Description: Percentage of subjects with parasite clearance on Day 1 (24 hours after first dose), Day 2 (48 hours after first dose), and Day 3 (72 hours after first dose).
Time Frame: Days 1, 2, and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Pyronaridine Artesunate: Subjects receive oral active-pyronaridine artesunate (tablet 180:60 mg) + chloroquine-placebo, once a day for 3 consecutive days (D0, 1, and 2).
  Posology was based on body weight ranges with subjects receiving 1 to 4 tablets depending on their body weight. The actual dose range covered by this regimen was 7.2:2.4 mg/kg to 13.8:4.6 mg/kg.
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 218 | 209
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 71.6 [65.6 to 77.5] | 30.6 [24.4 to 36.9]
  Clearance rate (%) at Day 2 (48h after first dose) | 99.5 [98.6 to 100.0] | 88.0 [83.6 to 92.4]
  Clearance rate (%) at Day 3 (72h after first dose) | 100.0 [100.0 to 100.0] | 96.7 [94.2 to 99.1]

6. Secondary Outcome: Percentage of Subjects With Fever Clearance on Days 1, 2, and 3
Description: Percentage of subjects with fever clearance on Day 1 (24 hours after first dose), Day 2 (48 hours after first dose), and Day 3 (72 hours after first dose).
Time Frame: Day 1, 2, and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 168 | 154
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 78.6 [72.4 to 84.8] | 58.4 [50.7 to 66.2]
  Clearance rate (%) at Day 2 (48h after first dose) | 89.9 [85.3 to 94.4] | 88.3 [83.2 to 93.4]
  Clearance rate (%) at Day 3 (72h after first dose) | 97.0 [94.5 to 99.6] | 97.4 [94.9 to 99.9]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events, including clinically significant laboratory results, ECG, vital signs or physical examination abnormalities.
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Population: Safety population consists of all randomized subjects who received any amount of study medication, subjects were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 228 | 228
Participants
  Nr subj. with ≥1 AE | 92 | 72
  Nr subj. with ≥1 treatment-related AE | 27 | 23
  Nr subj. with ≥1 SAE | 2 | 0
  Nr subj. with ≥1 treatment-related SAE | 0 | 0
  Nr subj. with ≥1 severe or life-threatening AE | 0 | 2
  Nr subj. with ≥1 AE leading to death | 0 | 0
  Nr subj. ≥1 AE leading to study drug discontinuation | 0 | 2
  Nr subj. with ≥1 AE leading to study withdrawal | 0 | 2

8. Other Pre Specified Outcome: Percentage of Subjects With PCR-corrected Cure Rate on Days 14, 21, and 28
Description: Cure on Days 14, 21, and 28 is defined as the absence of P. vivax parasitaemia on Days 14, 21, and 28 irrespective of temperature (axillary, oral, tympanic, rectal) without previously meeting any of the criteria of treatment failure throughout the follow-up period.
Time Frame: Day 14, 21, and 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 216 | 200
percentage of subjects
  Cure rate (%) at Day 14 | 100.0 [98.3 to 100.0] | 99.5 [97.2 to 100.0]
  Cure rate (%) at Day 21: number analyzed (Participants) | 212 | 198
  Cure rate (%) at Day 21 | 100.0 [98.3 to 100.0] | 99.5 [97.2 to 100.0]
  Cure rate (%) at Day 28: number analyzed (Participants) | 206 | 194
  Cure rate (%) at Day 28 | 98.1 [95.1 to 99.4] | 97.9 [94.8 to 99.4]

9. Other Pre Specified Outcome: Percentage of Subjects With Crude and PCR-corrected Cure Rate on Day 42
Description: Cure on Day 42 is defined as the absence of P. vivax parasitaemia on Day 42 irrespective of temperature (axillary, oral, tympanic, rectal) without previously meeting any of the criteria of treatment failure throughout the follow-up period.
Time Frame: Day 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine Artesunate | Chloroquine
Number analyzed (Participants) | 216 | 200
percentage of subjects
  Crude cure rate (%): number analyzed (Participants) | 199 | 190
  Crude cure rate (%) | 95.5 [91.6 to 97.9] | 92.1 [87.3 to 95.5]
  PCR-corrected cure rate (%): number analyzed (Participants) | 201 | 188
  PCR-corrected cure rate (%) | 95.0 [91.0 to 97.6] | 94.1 [89.8 to 97.0]

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Arm/Group | Pyronaridine Artesunate | Chloroquine
All-Cause Mortality (participants affected / at risk) | 2/228 | 0/228
Serious Adverse Events (participants affected / at risk) | 2/228 | 0/228
Other Adverse Events (participants affected / at risk) | 90/228 | 72/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine Artesunate (N=228) | Chloroquine (N=228)
Pyrexia (General disorders) | 1 (1) | 0 (0) — Prolonged hospitalisation due to fever
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0) — Hospitalisation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine Artesunate (N=228) | Chloroquine (N=228)
Fatigue (General disorders) | 12 (12) | 11 (11)
Nasopharyngitis (Infections and infestations) | 13 (15) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 19 (19) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 30 (30) | 21 (22)
Headache (Nervous system disorders) | 45 (52) | 34 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No